CLINICAL TRIAL: NCT03852108
Title: Impact of a Procedure With Socio-aesthetic Care on Anxiety and Pain Scale in the Early Rest of Pulmonary Transplant.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique Hopitaux De Marseille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2018-33; IDRCB (Other: 2018-A01968-47)
Record Dates: First submitted 2019-02-01; First posted 2019-02-22 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Pulmonary Transplant
MeSH Terms: interventions — Patient Comfort

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group comfort care (Experimental): Socio-aesthetic care
  Interventions: Other: Comfort Care
- Group control (No Intervention): Conventional care

INTERVENTIONS:
Other: Comfort Care — Face, Hand and body care for 15 to 45 minutes
  Arms: Group comfort care

SUMMARY:
Pulmonary transplant is a valid therapy and now accept in some case of respiratory disease at final state of their evolution in selected patients according to morbidity associated. This exceptionnal procedure (+/- 350 patients per year) brings benefits in terms of survival and quality of life but stay nevertheless, an experience very gruelling, anxiogenic and painful with sometimes extend hospitalizations in intensive care and then in pneumology unit.

Transplant can generate several complications like infection or rejection which can be fatal. The rate of death a year after the transplant is around 27% and whom 5 years after is around 48% according Biomedicine Agency, 2016) It's also mar of physical consequences (pain, scrars) specific to this act and expose the patient to several psychologic disruptions (decrease of body reflect, difficulty to accept organ of an other person...) So post transplant period is a painful and frightening moment. However, fear is not only sensory, it's also an affective side involving unpleasant feelings, fear and anxiety. It's a subjective and personnal experience influenced by the culture, context and other psychologic variables.

The collateral effects of transplantation could be controlled through additionnal diverse comfort cares but no care protocoles can be validated, especially because of multiple confounding individuals factors.

Recent studies showed that socio-aesthetic care allow an improvment of pain perception after cardiac surgery or oncology treatment.

The investigators propose to evaluate by a randomized controlled study the effect of comfort care of socio-aesthetic type on anxiety and pain in the aftermath of a pulmonary transplant.

In their hypothese, comfort care as socio-aethetic (body care, massage, manicure, corrective make up) could bring a personnalized answer to these patients, adapting to their complaint and waiting. It could ease the pain, anxiety, decrease level of corrective care and their side effects.

In their study, socio-aesthetic care will be done by therapist with 15 years of experience and working since 2003 in the oncology unit at la Timone Hospital and since 2009 to psychiatry unit to la Conception Hospital

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* patient transfered in Respiratory Unit (Hôpital Nord, APHM) immediate following lung transplant
* Person affiliated with a social security system

Exclusion Criteria:

* Patient refusing post transplant following until 6 months
* History of skin allergy
* Persons deprived of their liberty, persons under guardianship or trusteeship, persons in an emergency
* Person not affiliated to a social security system or not entitled to

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2019-02-05 (Actual); Primary Completion 2021-02-05 (Actual); Study Completion 2023-08-09 (Actual)

PRIMARY OUTCOMES:
Significant change of anxiety | Day 1, Day 7, Day 14, Day 21, Month 3, Month 6
  Anxiety will be measured by STAI-Y (State Trait Anxiety Inventory)
Significant change of pain | Day 1, Day 7, Day 14, Day 21, Month 3, Month 6
  Pain will be measured by the Visual Analogue Scale of pain. "no pain" to "maximum pain imaginable"

CONTACTS AND LOCATIONS:
Locations (1):
- Assistance Publique des Hôpitaux de Marseille, Marseille, France